CLINICAL TRIAL: NCT03130660
Title: Short Versus Long Axis Ultrasound Guided Approach for Internal Jugular Vein Cannulations: A Prospective Randomised Controlled Trial.
Brief Title: Short Versus Long Axis Ultrasound Guided Approach for Internal Jugular Vein Cannulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Medical Sciences and SUM Hospital (Other)
Responsible Party: Principal Investigator, Shakti Bedanta Mishra, Associate Professor, Institute of Medical Sciences and SUM Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DMR/IMS.SH/SOA/170022
Record Dates: First submitted 2017-04-22; First posted 2017-04-26 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Ultrasonography; Central Line Complication
Keywords: central line; Central Line Complication
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: patient to be randomized to two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Axis Ultrasonography (Experimental): one person does both ultrasound and line insertion
  Interventions: Device: Ultrasonography
- Long Axis Ultrasonography (Experimental): one person does ultrasound and another inserts the central line
  Interventions: Device: Ultrasonography

INTERVENTIONS:
Device: Ultrasonography — Ultrasound guidance for central line

SUMMARY:
We plan to compare single person short axis view with two person long axis view

DETAILED DESCRIPTION:
Introduction: The guidelines for the use of bedside ultrasonography in the evaluation of critically ill patients published by the society of critical care medicine recommends short-axis view be used during insertion of central venous catheter (CVC) in internal jugular vein (IJV) to improve success rate1. The long axis view is considered better for cannulations as it helps in preventing posterior wall puncture but in the trials it has been found to be inconvenient for a single user2,3. We hypothesise that if two persons perform long axis cannulations i.e. one person will image the vein while the other punctures it will be equally convenient to single person doing the cannulations in short axis. The advantage we expect to see is lesser complications in long axis group.

Methodology:

Inclusion criteria: Any patient getting admitted to ICU and requiring central venous cannulations.

Exclusion: Lack of consent. Randomization: At a 1:1 ratio, to be achieved using a computer-generated random number sequence for 100 consecutive subjects Study intervention: Eligible patients will be randomized to a short-axis or long axis technique for ultrasound guided IJV cannulations. Ultrasound guidance will be performed dynamically using a single-operator technique for short axis and double operator technique for long axis view. Cannulations and USG is to be carried out by 2 trained Anaesthesiologists.

Definition:

1. Insertion time: Time taken from 1st puncture of skin to insertion of guide wire into the vein.
2. Total Procedure time: Time from when Ultrasound scan was started to complete suturing of the CVC line.
3. Number of needle sticks: Number of time punctures were done in the skin. Complications were noted as hematoma formation, posterior wall puncture, arterial puncture, extravasations of blood and pneumothorax.

All the times are to be noted by a bedside nurse who is not involved in the trial or knows the study hypothesis.

Statistical Analysis: An intention-to-treat analysis was performed. Insertion time, overall procedure time and number of needle sticks, and will be compared using Mann-Whitney U tests. The success rate and complication rate will be compared using Fisher exact tests. All statistical analyses will be performed with SPSS 20.0

ELIGIBILITY:
Inclusion Criteria:

* Any patient getting admitted to ICU and requiring central venous cannulations.

Exclusion Criteria:

* Lack of consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
time to insertion | 15 minutes
  time from skin puncture to insertion of guidewire

SECONDARY OUTCOMES:
Total Procedure time | 15 minutes
  Time from when Ultrasound scan was started to complete suturing of the CVC line.
Number of needle sticks | 15 minutes
  Number of time punctures were done in the skin
Complications | 48 hours
  hematoma formation, posterior wall puncture, arterial puncture, extravasations of blood and pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rath, MD, Study Director — IMS and Sum hospital
Locations (1):
- IMS and SUM Hospital, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: Undecided
We havent decided yet